CLINICAL TRIAL: NCT03529851
Title: Feasibility of a Web-based Patient Reported Outcome Symptom Monitoring Application in Danish Lung Cancer Patients - a Pilot Study
Brief Title: Feasibility of a Web-based Patient Reported Outcome Symptom Monitoring Application in Danish Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: Danish Cancer Society (Other); Danish Lung Cancer Group (Other)
Responsible Party: Principal Investigator, Rasmus Blechingberg Friis, MD, Principal Investigator, Regional Hospital West Jutland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHWJutland
Record Dates: First submitted 2018-04-24; First posted 2018-05-18 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer Stage IV
Keywords: Patient reported outcomes; Symptom monitoring; Follow-up
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO intervention (Experimental): Patients included will weekly fill in a 12 item questionaire via the internet during the 3 week study period.
  Interventions: Other: Weekly questionnaires

INTERVENTIONS:
Other: Weekly questionnaires — In case of alarming symptoms reported in the questionnaire, an alert is automatically sent to the hospital. The clinicians will contact the patient, confirm the symptoms and intervene according to standard practice.

SUMMARY:
The trial is a pilot study prior to a following phase III trial and is designed to test the feasibility, acceptability and technical usability of supplementary web-based follow-up in lung cancer via a patient-reported outcome application.

DETAILED DESCRIPTION:
This pilot study will test if the use of AmbuFlex (a generic on-line system for self-recorded patient reported outcomes) is feasible for a following randomized trial (PRO-WIDE trial - Patient Reported Outcomes used for Weekly Internet-based DEtection of progressive disease in lung cancer; a randomized controlled trial). The RCT (randomized controlled trial) will test if weekly supplementary internet-based self-monitoring of 12 core symptoms can increase survival in Danish lung cancer patients during follow-up or maintenance treatment. A threshold mechanism will automatically send an alert to the hospital in case of alarming symptoms and the patient will be contacted by the clinicians.

In the pilot study, initial interviews with 7-10 patients will explore possible missing items and conceptual issues in the questionnaire. Based on the results an adjustment of the questionnaire will be considered.

Then the system including the alert trigger mechanism will be tested on 20 patients in medical antineoplastic treatment for three consecutive weeks. Acceptability, usability and relevance will be evaluated by a questionnaire at the end of the study period. Inclusion-rate, number of alerts per completed questionnaire and time usage of alert-management will be registered. For final evaluation, interviews with two nurses and two doctors will be made at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV lung cancer in palliative treatment with 3 weeks treatment intervals and next planned attendance at the hospital after 3 weeks.
2. Access to internet connection
3. Performance status ≤ 2
4. Patient has given his/her written informed consent

Exclusion Criteria:

1. Persons deprived of liberty or under guardianship or curators
2. Dementia, mental alteration or psychiatric disease that can compromise informed consent from the patient and / or adherence to the protocol and the monitoring of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Techincal feasibility, acceptability and usability of the PRO system for patients | 3 weeks
  Measured by an evaluation questionnaire at the end of the pilot study categorized according to the specified topics with 5 response items for each question. All responses will be presented in a comprehensive chart.
Inclusion rate | 3 weeks
  Number of included patients per screened patients Reasons for non-participation
Time usage per day on approval and handling alerts | 3 weeks
  Minutes spent per alert Minutes spent per telephone call
Barriers for implementation of the PRO system according to the clinical staff | 3 weeks
  Identified through interviews with 2 nurses and 2 MDs after the study period
Exploration of possible missing items and conceptual issues in the questionnaire. | 3 weeks
  Identified through interviews with 7-10 patients prior to the pilot study.
Alert-rate | 3 weeks
  Number of alerts sent to the hospital per questionnaires completed

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Friis, MD, Principal Investigator — Department of Oncology, Regional Hospital West Jutland
Locations (1):
- Department of oncology, Regional Hospital West Jutland, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friis RB, Hjollund NH, Mejdahl CT, Pappot H, Skuladottir H. Electronic symptom monitoring in patients with metastatic lung cancer: a feasibility study. BMJ Open. 2020 Jun 17;10(6):e035673. doi: 10.1136/bmjopen-2019-035673. PMID 32554725